CLINICAL TRIAL: NCT03581344
Title: Evaluation of the Interval Between Chemoradiotherapy and Surgery on Locally Advanced Rectal Cancer Response:a Multicentric Randomized Phase III Study
Brief Title: BReak Interval Delayed Surgery for Gastrointestinal Extraperitoneal Rectal Cancer
Acronym: BRIDGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, GAMBACORTA MARIA ANTONIETTA, Professor, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1908
Record Dates: First submitted 2018-06-14; First posted 2018-07-10 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Rectal Cancer
Keywords: Conservative Treatment; Neoadjuvant Therapy; Radiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The Patients included in the study will undergo a chemoradiotherapy neoadjuvant treatment.
  Patients will undergo a clinical-instrumental restaging at 7-8 weeks and will be randomized in two groups in case of major or complete response:
  1. Surgery 9-11 weeks after the end of neoadjuvant treatment
  2. Second clinical and instrumental re-evaluation after 11-12 weeks and then surgery 13-16 weeks after the end of chemoradiotherapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Patients undergoing surgery 9-11 weeks after the end of chemoradiotherapy, whose major/complete response has to be assessed with clinical-instrumental exams to be performed 7-8 weeks after the end of chemoradiotherapy.
- Experimental arm (Experimental): Patients undergoing surgery 13-16 weeks after the end of chemoradiotherapy, (length of surgical interval ) showing a major/complete response at the clinical-instrumental exams to be performed 7-8 weeks after the end of chemoradiotherapy. These patients will undergo a repetition of re-staging (a second clinical and instrumental re-evaluation after 11-12 weeks and then surgery 13-16 weeks after the end of chemoradiotherapy.)
  Interventions: Diagnostic Test: Repetition of Re-staging

INTERVENTIONS:
Diagnostic Test: Repetition of Re-staging — Second clinical and instrumental re-evaluation after 11-12 weeks and then surgery 13-16 weeks after the end of chemoradiotherapy if major or complete response at 7-8 weeks
  Arms: Experimental arm

SUMMARY:
This is a randomized multicentric clinical trial in patients affected by resectable rectal cancer, cT2N1-2, cT3N0-2, MRF -, aiming to evaluate the impact of the interval between chemoradiotherapy and surgery on the pathological response.

Patients will undergo a neoadjuvant chemoradiotherapy treatment and those achieving a major or complete clinical and instrumental response will then be randomized and submitted to surgery with two options: the first group will be operated after an interval of 9-11 weeks, while the second will undergo surgery at 13-16 weeks, after a further clinical and instrumental re-evaluation 11-12 weeks after the end of chemoradiotherapy.

DETAILED DESCRIPTION:
The proposed study is a randomized multicentric phase III study. The Patients included in the study will undergo a chemoradiotherapy neoadjuvant treatment.

Patients will undergo a clinical-instrumental restaging at 7-8 weeks and will be randomized in two groups in case of major or complete response:

1. Surgery 9-11 weeks after the end of neoadjuvant treatment
2. Second clinical and instrumental re-evaluation after 11-12 weeks and then surgery 13-16 weeks after the end of chemoradiotherapy.

Only patients who underwent preoperative chemoradiotherapy and achieved a complete or major response at the clinical-instrumental restaging 7-8 weeks after the end of neoadjuvant treatment will be included in the study.

The control arm of the BRIDGE-1 study is represented by patients undergoing surgery 9-11 weeks after the end of chemoradiotherapy, whose major/complete response has to be assessed with clinical-instrumental exams to be performed 7-8 weeks after the end of chemoradiotherapy.

The experimental arm of the the BRIDGE-1 study is represented by patients undergoing surgery 13-16 weeks after the end of chemoradiotherapy, showing a major/complete response at the clinical-instrumental exams to be performed 7-8 weeks after the end of chemoradiotherapy. These patients will undergo a new clinical and instrumental evaluation, 11-12 weeks after the end of neoadjuvant chemoradiotherapy treatment, prior to be submitted to the delayed surgical procedure.

Patients will be recruited in the two different arms, according to a randomized assignment, realized through an electronic table, in order to assure the efficacy of this study. Patients will be divided according to gender, age, stage and tumour site (low, medium and high) in each centre.

When a patient will be assigned to a specific arm, the randomization procedure will recruit a similar patient in the other arm.

CLINICAL STAGING AND RESTAGING EVALUATION TNM clinical and pathological stages are reported according to the American Joint Committee on Cancer 7th Edition, adenocarcinoma histological grading according to WHO classification.

Staging and baseline clinical evaluation

1. Patient history
2. Digital rectal examination
3. Recto-colonoscopy + biopsy (in case of impossibility to perform colonoscopy due to stenosing lesion, rectoscopy + biopsy and double-contrast barium enema or colon CT or colonoscopy within 6 months from surgery are suggested)
4. Pelvic MRI for loco-regional staging
5. CT of the thorax and abdomen for distant metastases staging
6. PET-CT (optional)
7. CEA test
8. Quality of Life (QoL) questionnaires compilation

Restaging at 7-8 weeks

1. Digital rectal examination
2. Pelvic MRI
3. PET-CT if performed during staging
4. Rectoscopy (in case of major/complete response)
5. CEA test
6. Quality of Life (QoL) questionnaires compilation

7.3 Restaging at 11-12 weeks (for patients randomized in the delayed surgery arm)

1. Digital rectal examination
2. Pelvic MRI
3. PET-CT if previously performed
4. Rectoscopy
5. CEA test

As secondary outcomes, acute and late toxicities, quality of life, bowel function, rectal continence and sexual activity will be evaluated in this study.

PREOPERATIVE CHEMORADIOTHERAPY TREATMENT Chemoradiotherapy treatment schedule considers a total radiotherapy dose of 55 Gy in 5 weeks, delivered with a 3D concomitant boost or Intensity Modulated Radiation Therapy (IMRT) Simultaneous Integrated Boost (SIB) technique.

Concomitant chemotherapy considers administration of Capecitabine for the whole radiotherapy course.

SURGICAL APPROACH Surgery will be performed according to standard techniques using the " open " approach, laparoscopic or robotic, according to surgeon's preference and including both anterior resection of the rectum and abdominoperineal rectal resection with mesorectal total excision (Total Mesorectal Excision, TME).

The possibility of sphincter salvage will be evaluated collectively by the members of the multidisciplinary team at the time of diagnosis, at first re-evaluation and in case of second re-evaluation.

PATHOLOGICAL EVALUATION Resected rectal specimens will undergo gross examination in order to macroscopically evaluate the status of the mesorectal margin.

After marking with indian ink the mesorectal margin, cutting axially the colorectal segment on its anti-mesorectal side and fixating it in formalin, transverse sections of the surgical specimen will be serially cut.

In case of macroscopic evidence of disease, sampling of the most infiltrated area and of the tumoral area with the minimum distance from the mesorectal margin, which will be included, will be performed.

In case of macroscopic absence or in the suspect of residual disease, the initial tumour site will be completely included in the specimen, localizing it from clinical reports with the potential aid of endoscopic tattoos and/or tissue alterations by the treatment (scar retraction or increase of tissue consistency).

In case of negative reports of the first histological sections, each inclusion will undergo three levels of histological section series.

The histopathological evaluation of the response to the therapy will be scored according to the following classifications: Mandard A.M., et al; Washington MK et al/College of American Pathologists; in presence of positive nodes, the Nottingham Rectal Cancer Prognostic Index (NRPI) score will also be used.

ADJUVANT CHEMOTHERAPY The protocol does not establish criteria for the administration of adjuvant systemic treatment.

The single center maintains the discretion to administer postoperative chemotherapy.

FOLLOW-UP The follow-up program recommended in the study is described in the national guidelines in effect.

Patients will undergo a clinical evaluation 1 month after surgery, every third month during the first year and then every sixth month up to the fifth year.

During follow-up visits the following tests will be performed and evaluated :

1. Physical examination and digital rectal exam ;
2. CEA and routine blood chemistry screen ;
3. Colonoscopy (at 1 year, if negative repeat after 3 years, if still negative repeat after 5 years) ;
4. Thoracic-abdominal-pelvic CT 3 months after surgery and then every sixth 6 month for the first 2 years, then annually (unless different clinical indication, i.e. suspicious lesions requiring short-term monitoring), in rotation with abdominal US ;
5. Complete abdominal US, each 6 months for the first 2 years, the annually (unless different clinical indication, i.e. suspicious lesions requiring short-term monitoring), in succession with Thoracic-abdominal-pelvic CT ;
6. Adverse events report (CTCAE v.04)
7. Quality of life (QoL) questionnaires to be filled during first follow up visits and then at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status 0-1
* Histological confirmation of Adenocarcinoma
* Rectal tumor localized within 12 cm from the internal anal sphincter (IAS)
* Clinical stage cT2N1-2, M0; cT3, N0-N2, M0 and MRF - , EMVI -
* Absence of major comorbidities contraindicating oncological treatments
* Major/complete clinical-instrumental response after CRT treatment
* Informed consent acquisition

Exclusion Criteria:

* cT4 and/or mesorectal fascia involvement (MRF+) and or EMVI +
* T localized at a distance > 12 cm from the internal anal sphincter (IAS)
* Presence of extramesorectal nodes
* Presence of distant metastases
* Pregnancy or breastfeeding status
* Diagnosis of tumor in other sites treated within the last five years, with the exception of basal cell skin carcinoma or in situ carcinoma of the cervix
* Absolute contraindication to pelvic radiotherapy, chemotherapy and/or surgery
* Contraindication to magnetic resonance imaging and/or endoscopy
* Informed consent absence
* Partial response, "no-change" or disease progression at restaging after 7-8 weeks from CRT end

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-09-17 (Estimated); Study Completion 2023-09-17 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) ypT0N0 | 9-16 weeks: surgery
  Absence of tumoral cells in the rectum and mesorectal nodes, examined by the pathologist
TRG (Tumor Regression Grade) | 9-16 weeks: surgery
  Histological assessment of the response of rectal cancer to neoadjuvant treatment

SECONDARY OUTCOMES:
Overall survival | 24-60 months
  The length of time from either the date of diagnosis that patients diagnosed with the disease are still alive
Disease free survival | 24-60 months
  The length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer
Local recurrence free survival | 24-60 months
  The length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of local recurrence
Metastasis free survival | 24-60 months
  The length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of distant metastasis
Concordance between major clinical response (ymCR) or complete clinical response (ycCR) at imaging and ypCR | 24-60 months
  Concordance between clinical-instrumental restaging and analysis of pathological specimen
Colostomy free survival | 24-60 months
  The length of time after primary treatment for a cancer ends that the patient survives without colostomy
Impact of therapy on bowel function | 24-60 months
  Evaluating impact of therapy on bowel function according to MSKCC questionary (Temple LK and al, Dis Colon Rectum 2005: 48: 1353-1365)
  The MSKCC Bowel Function questionnaire is a selfadministered psychometric instrument designed to assess bowel function in patients who undergo sphincterpreserving surgery for rectal cancer. The questionnaire includes 18 items involving three subscales (frequency, dietary and urgency/soilage), four individual items of clinical significance (Q4: incomplete emptying after a bowel movement, Q6: a second bowel movement within 15 min, Q7: knowing difference between gas and bowel movements, Q12: unable to control the passage of flatus) and one total score that is obtained by summing all 18 items.
Impact of therapy on fecal continence | 24-60 months
  Evaluating impact of therapy on fecal incontinence according to Fecal Incontinence Quality of Life Instrument (Rockwood et al., Dis Colon Rectum. 2000 Jan;43(1):9-16; discussion 16-7).
  Total of 29 items; these items form four scales: Lifestyle (10 items), Coping/Behavior (9 items), Depression/Self-Perception (7 items), and Embarrassment. (3 items).
  Scales range from 1 to 5, with a 1 indicating a lower functional status of quality of life. Scale scores are the average (mean) response to all items in the scale Scale 1. Lifestyle, ten items: Q2a Q2b Q2c Q2d Q2e Q2g Q2h Q3b Q31 Q3m Scale 2. Coping/Behavior, nine items: Q2f Q2i Q2j Q2k Q2m Q3d Q3h Q3j Q3n Scale 3. Depression/Self Perception, seven items: Q1 Q3d Q3f Q3g Q3i Q3k Q4, (Question 1 is reverse coded.) Scale 4. Embarrassment, three items: Q21 Q3a Q3e
Impact of therapy on sexual activity | 24-60 months
  Evaluating impact of therapy on fecal incontinence according to European Organisation for the Research and Treatment of Cancer (EORTC) QLQ - CR29 It is composed of 29 items that evaluate symptoms (gastrointestinal, urinary, pain and others) and functional areas (sexual, body image and others) that are associated with colorectal cancer and its treatments. There are separate scales for patients with or without stoma (which can be compared) and separate items to evaluate sexual function for men and women. The questionnaire has a Likert scale of four response categories.
Impact of therapy on quality of life (QoL) | 24-60 months
  Evaluating impact of therapy on fecal incontinence according to EORTC QLQ-C30 It is composed of both multi-item scales and single-item measures. These include 5 functional scales, 3 symptom scales, a global health status / QoL scale, and 6 single items. Each of the multi-item scales includes a different set of items. All of the scales and single-item measures range in score from 0 to 100.
  Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
  For scoring these scales:
  1. Estimate the average of the items that contribute to the scale; this is the raw score.
  2. Use a linear transformation to standardise the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione policlinico universitario a. gemelli IRCCS, Rome, Italy

REFERENCES:
- [Derived] Chiloiro G, Meldolesi E, Corvari B, Romano A, Barbaro B, Coco C, Crucitti A, Genovesi D, Lupattelli M, Mantello G, Menghi R, Falchetto Osti M, Persiani R, Petruzziello L, Ricci R, Sofo L, Valentini C, De Paoli A, Valentini V, Antonietta Gambacorta M. BRIDGE -1 TRIAL: BReak Interval Delayed surgery for Gastrointestinal Extraperitoneal rectal cancer, a multicentric phase III randomized trial. Clin Transl Radiat Oncol. 2022 Mar 8;34:30-36. doi: 10.1016/j.ctro.2022.03.002. eCollection 2022 May. PMID 35340685